CLINICAL TRIAL: NCT03257995
Title: A Randomized, Double-blind, Placebo-controlled, Three-period Cross-over Study to Assess the Pharmacodynamics, Safety, Tolerability, and Pharmacokinetics of Two Orally Inhaled Indacaterol Salts (Maleate and Acetate) Delivered Via the Concept1 Inhalation Device in Patients With Asthma
Brief Title: Pharmacodynamics, Safety, Tolerability, and Pharmacokinetics of Two Orally Inhaled Indacaterol Salts in Adult Subjects With Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVM149B2203
Record Dates: First submitted 2017-06-06; First posted 2017-08-22 (Actual); Results first posted 2019-03-29 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Asthma
Keywords: asthma, asthma attack, difficulty breathing, bronchial diseases, lung, lung diseases, inhaled drugs, bronchodilator, inhaled corticosteriod
MeSH Terms: conditions — Asthma; Dyspnea; Bronchial Diseases; Lung Diseases | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): A-B-C
  Interventions: Drug: Indacaterol maleate; Drug: Indacaterol acetate; Drug: Placebo
- Sequence 2 (Experimental): B-C-A
  Interventions: Drug: Indacaterol maleate; Drug: Indacaterol acetate; Drug: Placebo
- Sequence 3 (Experimental): C-A-B
  Interventions: Drug: Indacaterol maleate; Drug: Indacaterol acetate; Drug: Placebo
- Sequence 4 (Experimental): A-C-B
  Interventions: Drug: Indacaterol maleate; Drug: Indacaterol acetate; Drug: Placebo
- Sequence 5 (Experimental): B-A-C
  Interventions: Drug: Indacaterol maleate; Drug: Indacaterol acetate; Drug: Placebo
- Sequence 6 (Experimental): C-B-A
  Interventions: Drug: Indacaterol maleate; Drug: Indacaterol acetate; Drug: Placebo

INTERVENTIONS:
Drug: Indacaterol maleate — 150 μg via Concept1 device
  Other Names: A
Drug: Indacaterol acetate — 150 μg via Concept1 device
  Other Names: B
Drug: Placebo — Capsule containing no active ingredients delivered via Concept1 device
  Other Names: C

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, three-period cross-over study in approximately 54 subjects with asthma.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, three-period cross-over study in asthma patients. The study will consist of a screening epoch, followed by a treatment epoch which consists of three treatment periods, and will conclude with an end of study epoch.

Each subject will be assigned to 1 of 6 treatment sequences and will sequentially receive the investigational products and placebo during the trial.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female patients aged ≥ 18 and above
* Patients with a documented physician diagnosis of asthma for a period of at least 1 year prior to screening and who additionally meet the following criteria:

Patients receiving daily treatment with an inhaled corticosteroid up to the maximum dose per day (as indicated in the package leaflet), on a stable regimen for at least 4 weeks prior to screening.

* Pre-bronchodilator FEV1 ≥ 50 % and ≤ 90% of the predicted normal value for the patient during screening.
* Patients who demonstrate an increase in FEV1 of ≥ 12% and ≥ 200 mL after administration of 400 μg salbutamol/360 μg albuterol (or equivalent dose) at screening.
* Subjects must weigh at least 50 kg at screening to participate in the study, and must have a body mass index (BMI) within the range of 18 to 40 kg/m2.

Key Exclusion Criteria:

-Contraindicated for treatment with, or having a history of reactions/ hypersensitivity to any of the following inhaled drugs, drugs of a similar class, or any component thereof: Sympathomimetic amines / adrenoceptor agonist agents Lactose or any of the other excipients of the study drug (including patients with history of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption)

* Patients who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 6 weeks of screening.
* Patients who have had a respiratory tract infection or asthma worsening within 4 weeks prior to screening.
* Patients with a history of chronic lung diseases other than asthma
* Patients who have a decline in PEF from the reference PEF (taken at screening) of ≥30% for 5 of 6 consecutive scheduled PEF readings (readings taken at morning and evening) during at least 3 days of screening epoch prior to randomization.
* Patients who require the use of ≥12 puffs / 24 hours of rescue medication for 48 hours (over two consecutive days) during screening prior to randomization.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Patients with Type I diabetes or uncontrolled Type II diabetes (HbA1c > 9%) at screening.
* Current smokers (urine cotinine > than the laboratory's lowest level of quantification (LoQ of 500 ng/mL or lower)) and patients who have smoked or inhaled tobacco products within the 6 month period prior to screening, or who have a smoking history of greater than 10 pack years (Note: 1 pack is equivalent to 20 cigarettes. 10 pack years = 1 pack /day x 10 yrs., or ½ pack/day x 20 yrs.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-01-17 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Skillman, New Jersey
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Medford, Oregon
  - Novartis Investigative Site, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Miller D, Vaidya S, Jauernig J, Ethell B, Wagner K, Radhakrishnan R, Tillmann HC. Lung function, pharmacokinetics, and tolerability of inhaled indacaterol maleate and acetate in asthma patients. Respir Res. 2020 Sep 23;21(1):248. doi: 10.1186/s12931-020-01501-1. PMID 32967685
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=438

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: indacaterol maleate 150 μg , indacaterol acetate 150 μg and matching placebo
- Sequence 2: indacaterol acetate 150 μg, matching placebo and indacaterol maleate 150 μg
- Sequence 3: Placebo, indacaterol maleate 150 μg and indacaterol acetate 150 μg
- Sequence 4: indacaterol maleate 150 μg, placebo, and indacaterol acetate 150 μg
- Sequence 5: indacaterol acetate 150 μg, indacaterol maleate 150 μg, and placebo
- Sequence 6: Placebo, indacaterol acetate 150 μg, indacaterol maleate 150 μg
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 9 | 9 | 9 | 9 | 9 | 9
Completed | 9 | 8 | 9 | 9 | 9 | 7
Not Completed | 0 | 1 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized to one of six treatment sequences
Arm/Group | All Participants
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1
Description: FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of forced exhalation. Treatment differences in trough FEV1 after 14 days of treatment between indacaterol maleate 150 μg and placebo, between indacaterol acetate 150 μg and placebo and indacaterol maleate and indacaterol acetate
Time Frame: Day 14 of each of the three treatment periods
Population: The PD analysis set included all patients with available PD parameter data who received any study drug and experienced no major protocol deviations with relevant impact on PD data
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Indacaterol Maleate: indacaterol maleate 150 μg via Breezhaler
- Indacaterol Acetate: indacaterol acetate 150 μg via Breezhaler
- Placebo: matching placebo capsules to indacaterol via Breezhaler
Arm/Group | Indacaterol Maleate | Indacaterol Acetate | Placebo
Number analyzed (Participants) | 51 | 52 | 53
Liters | 2.4173 (0.78214) | 2.3774 (0.77679) | 2.2191 (0.72350)
Statistical Analysis 1: Comparison: Indacaterol Maleate vs Placebo; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1861, 95% CI 2-sided [0.1293 to 0.2429]
Statistical Analysis 2: Comparison: Indacaterol Acetate vs Placebo; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1463, 95% CI 2-sided [0.0898 to 0.2029]
Statistical Analysis 3: Comparison: Indacaterol Maleate vs Indacaterol Acetate; Test type: Other; ANOVA; Mean Difference (Final Values) = -0.0398, 95% CI 2-sided [-0.0942 to 0.0147]

2. Secondary Outcome: Pharmacokinetics AUC 0-24hours at Steady State
Description: AUC 0-24hours of plasma concentrations of indacaterol maleate and indacaterol acetate at steady state.The area under the concentrations-time curve (AUC0-24) was calculated with the measured data points from the time of administration up to 24 h after administration by the trapezoidal formula. The concentration-time curve is the result of time points of blood sampling and its measured concentration in the blood samplings
Time Frame: Day 14 of each of the three treatment periods
Population: The PK analysis set included all patients with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study drug and experienced no major protocol deviations with relevant impact on PK data.
Measure: Mean (Standard Deviation); unit: h*pg/mL
Groups:
- Indacaterol Maleate 150 µg: indacaterol maleate 150 μg via Breezhaler
- Indacaterol Acetate 150 µg: indacaterol acetate 150 μg via Breezhaler
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg
Number analyzed (Participants) | 51 | 52
h*pg/mL | 2300 (732) | 2050 (636)

3. Secondary Outcome: The Maximum Concentration (Cmax) at Steady State (ss)
Description: Maximal plasma concentrations of indacaterol maleate and indacaterol acetate at steady state. The maximum concentration (Cmax) were obtained directly from the measured concentration-time curves. The concentration-time curve is the result of time points of blood sampling and its measured concentration in the blood samplings.
Time Frame: Day 14 of each of the three treatment periods
Population: as for outcome 2
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg
Number analyzed (Participants) | 51 | 52
pg/mL | 249 [126 to 443] | 224 [84.9 to 426]

4. Secondary Outcome: Time of Maximal Plasma Concentration (Tmax) at Steady State
Description: Time of maximal plasma concentration of indacaterol maleate and indacaterol acetate at steady state. Time to reach the maximum concentration after administration. In this analysis Tmax will be reported using blood samples taken on Days 14
Time Frame: Day 14 of each of the three treatment periods
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg
Number analyzed (Participants) | 51 | 52
h | 0.250 [0.183 to 0.850] | 0.467 [0.183 to 1.00]

5. Secondary Outcome: The Lowest Plasma (or Serum or Blood) Concentration (Cmin) at Steady State
Description: The lowest plasma (or serum or blood) concentration observed during a dosing interval at steady state. Only summary statistics was provided.
Time Frame: Day 14 of each of the three treatment periods
Population: as for outcome 2
Measure: Median (Full Range); unit: pg/mL
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg
Number analyzed (Participants) | 51 | 52
pg/mL | 56 [14.5 to 126] | 52.3 [9.03 to 106]

6. Secondary Outcome: Relative Bioavailability (Frel) of Indacaterol Acetate and Indacaterol Maleate
Description: Relative bioavailability will be determined for AUC0-24h,ss and Cmax,ss comparing systemic exposure of indacaterol acetate and indacaterol maleate.
Time Frame: Day 14
Population: The PK analysis set included all patients with at least one available valid (i.e. not flagged for exclusion) PK concentration measurement, who received any study drug and experienced no major protocol deviations with relevant impact on PK data. Only summary statistics for relative bioavailability was provided.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- Indacaterol Maleate / Indacaterol Acetate: Relative bioavailability of indacaterol acetate compared to indacaterol maleate (Frel) AUC0-24h,ss
- Indacaterol Acetate 150 µg: Relative bioavailability of indacaterol acetate compared to indacaterol maleate (Frel) Cmax,ss
Arm/Group | Indacaterol Maleate / Indacaterol Acetate | Indacaterol Acetate 150 µg
Number analyzed (Participants) | 43 | 45
Ratio | 0.912 (0.201) | 0.910 (0.242)

7. Secondary Outcome: Time to Peak FEV1 on Day 14
Description: The differences in median time to peak FEV1 (h) between indacaterol maleate 150 µg and placebo
Time Frame: Day 14 of each of the three treatment periods
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: h
Arm/Group | Indacaterol Maleate | Indacaterol Acetate | Placebo
Number analyzed (Participants) | 51 | 51 | 51
h | -0.02 [-0.83 to 0.33] | -0.02 [-0.82 to 0.51] | 0.00 [-0.50 to 0.73]
Statistical Analysis 1: Comparison: Indacaterol Maleate; Test type: Other; p = 0.823, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.02, 95% CI 2-sided [-0.83 to 0.33]
Statistical Analysis 2: Comparison: Indacaterol Acetate; Test type: Other; p = 0.801, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -0.02, 95% CI 2-sided [-0.82 to 0.51]
Statistical Analysis 3: Comparison: Placebo; Test type: Other; p = 0.984, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.00, 95% CI 2-sided [-0.50 to 0.73]

8. Secondary Outcome: Bronchodilator Effect of Indacaterol Salts Compared to Placebo Measured by Forced Expiratory Volume in 1 Second (FEV1) at All Timepoints
Description: Bronchodilator effect of indacaterol salts compared to placebo in terms of FEV1. Day 14, FEV1 was measured at 24hours post dose
Time Frame: Day 14 of each of the three treatment periods at 5, 15, 30m, 1 2, 3, 4, 8, 12, 23hour.15min and 23hour.45min
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liter
Arm/Group | Indacaterol Maleate | Indacaterol Acetate | Placebo
Number analyzed (Participants) | 51 | 52 | 53
Liter
  5 min: number analyzed (Participants) | 51 | 52 | 50
  5 min | 2.4795 [2.2575 to 2.7014] | 2.4813 [2.2595 to 2.7031] | 2.2617 [2.0398 to 2.4837]
  15 min: number analyzed (Participants) | 51 | 49 | 51
  15 min | 2.5005 [2.2786 to 2.7224] | 2.4965 [2.2746 to 2.7184] | 2.2282 [2.0062 to 2.4501]
  30 min: number analyzed (Participants) | 51 | 51 | 51
  30 min | 2.5204 [2.2985 to 2.7424] | 2.5047 [2.2829 to 2.7265] | 2.2475 [2.0255 to 2.4694]
  1 hour: number analyzed (Participants) | 51 | 52 | 51
  1 hour | 2.5279 [2.3060 to 2.7498] | 2.5018 [2.2800 to 2.7236] | 2.2670 [2.0451 to 2.4889]
  2 hour: number analyzed (Participants) | 51 | 51 | 51
  2 hour | 2.5286 [2.3067 to 2.7505] | 2.5338 [2.3120 to 2.7556] | 2.2792 [2.0573 to 2.5011]
  4 hour: number analyzed (Participants) | 51 | 51 | 50
  4 hour | 2.5054 [2.2835 to 2.7273] | 2.5103 [2.2885 to 2.7321] | 2.2781 [2.0561 to 2.5001]
  8 hour: number analyzed (Participants) | 49 | 51 | 49
  8 hour | 2.4668 [2.2448 to 2.6888] | 2.4596 [2.2378 to 2.6814] | 2.2272 [2.0052 to 2.4492]
  12 hour: number analyzed (Participants) | 49 | 51 | 48
  12 hour | 2.4222 [2.2002 to 2.6442] | 2.3836 [2.1618 to 2.6054] | 2.1779 [1.9558 to 2.3999]
  23 hour 15 min: number analyzed (Participants) | 47 | 50 | 41
  23 hour 15 min | 2.4678 [2.2457 to 2.6899] | 2.4022 [2.1804 to 2.6241] | 2.2398 [2.0173 to 2.4622]
  23 hour 45 min: number analyzed (Participants) | 47 | 50 | 41
  23 hour 45 min | 2.4585 [2.2364 to 2.6806] | 2.4424 [2.2205 to 2.6642] | 2.2631 [2.0407 to 2.4856]
Statistical Analysis 1: Comparison: Indacaterol Maleate vs Placebo; at 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2177, 95% CI 2-sided [0.1482 to 0.2872]
Statistical Analysis 2: Comparison: Indacaterol Maleate vs Placebo; 15min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2724, 95% CI 2-sided [0.2030 to 0.3417]
Statistical Analysis 3: Comparison: Indacaterol Maleate vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2730, 95% CI 2-sided [0.2036 to 0.3423]
Statistical Analysis 4: Comparison: Indacaterol Maleate vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2609, 95% CI 2-sided [0.1915 to 0.3302]
Statistical Analysis 5: Comparison: Indacaterol Maleate vs Placebo; 2 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2494, 95% CI 2-sided [0.1800 to 0.3188]
Statistical Analysis 6: Comparison: Indacaterol Maleate vs Placebo; 4 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2273, 95% CI 2-sided [0.1578 to 0.2968]
Statistical Analysis 7: Comparison: Indacaterol Maleate vs Placebo; 8 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2396, 95% CI 2-sided [0.1697 to 0.3096]
Statistical Analysis 8: Comparison: Indacaterol Maleate vs Placebo; 12 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2443, 95% CI 2-sided [0.1742 to 0.3144]
Statistical Analysis 9: Comparison: Indacaterol Maleate vs Placebo; 23 hour 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2280, 95% CI 2-sided [0.1563 to 0.2997]
Statistical Analysis 10: Comparison: Indacaterol Maleate vs Placebo; 23 hour 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1954, 95% CI 2-sided [0.1237 to 0.2671]
Statistical Analysis 11: Comparison: Indacaterol Acetate vs Placebo; 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2195, 95% CI 2-sided [0.1502 to 0.2889]
Statistical Analysis 12: Comparison: Indacaterol Acetate vs Placebo; 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2684, 95% CI 2-sided [0.1988 to 0.3380]
Statistical Analysis 13: Comparison: Indacaterol Acetate vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2572, 95% CI 2-sided [0.1879 to 0.3266]
Statistical Analysis 14: Comparison: Indacaterol Acetate vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2348, 95% CI 2-sided [0.1656 to 0.3040]
Statistical Analysis 15: Comparison: Indacaterol Acetate vs Placebo; 2 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2546, 95% CI 2-sided [0.1852 to 0.3239]
Statistical Analysis 16: Comparison: Indacaterol Acetate vs Placebo; 4 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2322, 95% CI 2-sided [0.1627 to 0.3017]
Statistical Analysis 17: Comparison: Indacaterol Acetate vs Placebo; 8 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2324, 95% CI 2-sided [0.1627 to 0.3020]
Statistical Analysis 18: Comparison: Indacaterol Acetate vs Placebo; 12 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2057, 95% CI 2-sided [0.1359 to 0.2755]
Statistical Analysis 19: Comparison: Indacaterol Acetate vs Placebo; 23 hour 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1625, 95% CI 2-sided [0.0912 to 0.2337]
Statistical Analysis 20: Comparison: Indacaterol Acetate vs Placebo; 23 hour 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1793, 95% CI 2-sided [0.1080 to 0.2505]

9. Secondary Outcome: Percent of Predicted Bronchodilator Effect of Indacaterol Salts Compared to Placebo Measured by FEV1 (% Predicted) at All Timepoints
Description: The FEV1 percent predicted expresses FEV1 as a percentage of the "predicted values" for participants of similar characteristics (height, age, sex, and sometimes race and weight). A positive change from baseline in FEV1 % predicted indicates improvement in lung function. FEV1 % predicted was assessed at each post dose time point after 14 days
Time Frame: Day 14 of each of the three treatment periods at 5, 15, 30m, 1 2, 3, 4, 8, 12, 23hour.15min and 23hour.45min
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of predicted
Arm/Group | Indacaterol Maleate | Indacaterol Acetate | Placebo
Number analyzed (Participants) | 51 | 52 | 53
Percent of predicted
  5 min: number analyzed (Participants) | 51 | 52 | 50
  5 min | 78.2 [74.7 to 81.7] | 78.2 [74.8 to 81.7] | 71.1 [67.7 to 74.6]
  15 min: number analyzed (Participants) | 51 | 49 | 51
  15 min | 78.7 [75.2 to 82.2] | 78.5 [75.0 to 82.0] | 70.2 [66.7 to 73.7]
  30 min: number analyzed (Participants) | 51 | 51 | 51
  30 min | 79.4 [75.9 to 82.9] | 78.9 [75.4 to 82.3] | 70.7 [67.3 to 74.2]
  1 hour: number analyzed (Participants) | 51 | 52 | 51
  1 hour | 79.5 [76.0 to 83.0] | 78.8 [75.3 to 82.3] | 71.4 [67.9 to 74.9]
  2 hours: number analyzed (Participants) | 51 | 51 | 51
  2 hours | 79.6 [76.1 to 83.1] | 79.8 [76.3 to 83.2] | 72.0 [68.5 to 75.5]
  4 hours: number analyzed (Participants) | 51 | 51 | 50
  4 hours | 78.8 [75.4 to 82.3] | 79.1 [75.6 to 82.5] | 71.8 [68.3 to 75.3]
  8 hours: number analyzed (Participants) | 49 | 51 | 49
  8 hours | 77.5 [74.0 to 81.0] | 77.5 [74.1 to 81.0] | 70.2 [66.7 to 73.6]
  12 hours: number analyzed (Participants) | 49 | 51 | 48
  12 hours | 76.2 [72.7 to 79.7] | 75.0 [71.5 to 78.5] | 68.6 [65.2 to 72.1]
  23 hours 15 min: number analyzed (Participants) | 47 | 50 | 41
  23 hours 15 min | 77.9 [74.5 to 81.4] | 76.1 [72.6 to 79.5] | 71.0 [67.5 to 74.5]
  23 hours 45 min: number analyzed (Participants) | 47 | 50 | 41
  23 hours 45 min | 77.8 [74.3 to 81.3] | 77.2 [73.7 to 80.7] | 71.4 [67.8 to 74.9]
Statistical Analysis 1: Comparison: Indacaterol Maleate vs Placebo; at 5 min; Test type: Other; p < .001, ANOVA; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [5.0 to 9.2]
Statistical Analysis 2: Comparison: Indacaterol Maleate vs Placebo; at 15 min; Test type: Other; p < .001, ANOVA; Mean Difference (Final Values) = 8.5, 95% CI 2-sided [6.4 to 10.6]
Statistical Analysis 3: Comparison: Indacaterol Maleate vs Placebo; at 30; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 8.6, 95% CI 2-sided [6.5 to 10.7]
Statistical Analysis 4: Comparison: Indacaterol Maleate vs Placebo; at 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 8.0, 95% CI 2-sided [6.0 to 10.1]
Statistical Analysis 5: Comparison: Indacaterol Maleate vs Placebo; at 2 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.6, 95% CI 2-sided [5.5 to 9.7]
Statistical Analysis 6: Comparison: Indacaterol Maleate vs Placebo; at 4 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [5.0 to 9.1]
Statistical Analysis 7: Comparison: Indacaterol Maleate vs Placebo; at 8 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [5.2 to 9.4]
Statistical Analysis 8: Comparison: Indacaterol Maleate vs Placebo; at 12 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.6, 95% CI 2-sided [5.5 to 9.7]
Statistical Analysis 9: Comparison: Indacaterol Maleate vs Placebo; at 23 hours 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.0, 95% CI 2-sided [4.8 to 9.1]
Statistical Analysis 10: Comparison: Indacaterol Maleate vs Placebo; at 23 hours 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [4.2 to 8.6]
Statistical Analysis 11: Comparison: Indacaterol Acetate vs Placebo; at 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.1, 95% CI 2-sided [5.0 to 9.2]
Statistical Analysis 12: Comparison: Indacaterol Acetate vs Placebo; at 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 8.3, 95% CI 2-sided [6.2 to 10.4]
Statistical Analysis 13: Comparison: Indacaterol Acetate vs Placebo; at 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 8.1, 95% CI 2-sided [6.0 to 10.2]
Statistical Analysis 14: Comparison: Indacaterol Acetate vs Placebo; at 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [5.3 to 9.4]
Statistical Analysis 15: Comparison: Indacaterol Acetate vs Placebo; at 2 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.8, 95% CI 2-sided [5.7 to 9.9]
Statistical Analysis 16: Comparison: Indacaterol Acetate vs Placebo; at 4 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.3, 95% CI 2-sided [5.2 to 9.4]
Statistical Analysis 17: Comparison: Indacaterol Acetate vs Placebo; at 8 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 7.4, 95% CI 2-sided [5.3 to 9.5]
Statistical Analysis 18: Comparison: Indacaterol Acetate vs Placebo; at 12 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [4.2 to 8.4]
Statistical Analysis 19: Comparison: Indacaterol Acetate vs Placebo; at 23 hours 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.1, 95% CI 2-sided [2.9 to 7.2]
Statistical Analysis 20: Comparison: Indacaterol Acetate vs Placebo; at 23 hours 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.9, 95% CI 2-sided [3.7 to 8.0]

10. Secondary Outcome: Bronchodilator Effect of Indacaterol Salts Compared to Placebo Measured by Forced Vital Capacity (FVC)
Description: Forced Vital Capacity is the amount of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was assessed by spirometry at each post dose time point after 14 days. A positive change from baseline in FVC indicates improvement in lung function.
Time Frame: Day 14 of each of the three treatment periods at at 5, 15, 30m, 1 2, 3, 4, 8, 12, 23hour.15min and 23hour.45min
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 51 | 52 | 53
liter
  5 min: number analyzed (Participants) | 51 | 50 | 50
  5 min | 3.5648 [3.2407 to 3.8890] | 3.5912 [3.2672 to 3.9152] | 3.3783 [3.0541 to 3.7024]
  15 min: number analyzed (Participants) | 51 | 49 | 51
  15 min | 3.5850 [3.2608 to 3.9091] | 3.5773 [3.2531 to 3.9015] | 3.3600 [3.0359 to 3.6842]
  30 min: number analyzed (Participants) | 51 | 51 | 51
  30 min | 3.6068 [3.2827 to 3.9310] | 3.6039 [3.2798 to 3.9279] | 3.3664 [3.0422 to 3.6905]
  1 hour: number analyzed (Participants) | 51 | 52 | 51
  1 hour | 3.5946 [3.2705 to 3.9188] | 3.5886 [3.2645 to 3.9126] | 3.3873 [3.0631 to 3.7114]
  2 hour: number analyzed (Participants) | 51 | 51 | 51
  2 hour | 3.5789 [3.2548 to 3.9031] | 3.5992 [3.2751 to 3.9233] | 3.3987 [3.0745 to 3.7228]
  4 hour: number analyzed (Participants) | 51 | 51 | 50
  4 hour | 3.5674 [3.2433 to 3.8916] | 3.5999 [3.2759 to 3.9240] | 3.4053 [3.0812 to 3.7295]
  8 hour: number analyzed (Participants) | 49 | 51 | 49
  8 hour | 3.5670 [3.2428 to 3.8913] | 3.5617 [3.2376 to 3.8858] | 3.3680 [3.0438 to 3.6922]
  12 hour: number analyzed (Participants) | 49 | 51 | 48
  12 hour | 3.4941 [3.1698 to 3.8183] | 3.4812 [3.1571 to 3.8053] | 3.3193 [2.9950 to 3.6436]
  23 hour 15 min: number analyzed (Participants) | 47 | 50 | 41
  23 hour 15 min | 3.6055 [3.2812 to 3.9298] | 3.5448 [3.2207 to 3.8689] | 3.4199 [3.0952 to 3.7446]
  23 hour 45 min: number analyzed (Participants) | 47 | 50 | 41
  23 hour 45 min | 3.5668 [3.2425 to 3.8912] | 3.5731 [3.2489 to 3.8972] | 3.4185 [3.0938 to 3.7431]
Statistical Analysis 1: Comparison: Indacaterol Maleate 150 µg vs Placebo; 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1866, 95% CI 2-sided [0.1121 to 0.2611]
Statistical Analysis 2: Comparison: Indacaterol Maleate 150 µg vs Placebo; 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2249, 95% CI 2-sided [0.1506 to 0.2992]
Statistical Analysis 3: Comparison: Indacaterol Maleate 150 µg vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2404, 95% CI 2-sided [0.1661 to 0.3148]
Statistical Analysis 4: Comparison: Indacaterol Maleate 150 µg vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2074, 95% CI 2-sided [0.1330 to 0.2817]
Statistical Analysis 5: Comparison: Indacaterol Maleate 150 µg vs Placebo; 2 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1802, 95% CI 2-sided [0.1059 to 0.2545]
Statistical Analysis 6: Comparison: Indacaterol Maleate 150 µg vs Placebo; 4 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1621, 95% CI 2-sided [0.0876 to 0.2366]
Statistical Analysis 7: Comparison: Indacaterol Maleate 150 µg vs Placebo; 8 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1990, 95% CI 2-sided [0.1239 to 0.2742]
Statistical Analysis 8: Comparison: Indacaterol Maleate 150 µg vs Placebo; 12 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1747, 95% CI 2-sided [0.0994 to 0.2501]
Statistical Analysis 9: Comparison: Indacaterol Maleate 150 µg vs Placebo; 23 hours 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1856, 95% CI 2-sided [0.1081 to 0.2631]
Statistical Analysis 10: Comparison: Indacaterol Maleate 150 µg vs Placebo; 23 hours 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1484, 95% CI 2-sided [0.0709 to 0.2259]
Statistical Analysis 11: Comparison: Indacaterol Acetate 150 µg vs Placebo; 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2130, 95% CI 2-sided [0.1386 to 0.2873]
Statistical Analysis 12: Comparison: Indacaterol Acetate 150 µg vs Placebo; 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2173, 95% CI 2-sided [0.1426 to 0.2920]
Statistical Analysis 13: Comparison: Indacaterol Acetate 150 µg vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2375, 95% CI 2-sided [0.1632 to 0.3118]
Statistical Analysis 14: Comparison: Indacaterol Acetate 150 µg vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2013, 95% CI 2-sided [0.1272 to 0.2754]
Statistical Analysis 15: Comparison: Indacaterol Acetate 150 µg vs Placebo; 2 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2005, 95% CI 2-sided [0.1262 to 0.2749]
Statistical Analysis 16: Comparison: Indacaterol Acetate 150 µg vs Placebo; 4 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1946, 95% CI 2-sided [0.1201 to 0.2691]
Statistical Analysis 17: Comparison: Indacaterol Acetate 150 µg vs Placebo; 8 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1937, 95% CI 2-sided [0.1190 to 0.2684]
Statistical Analysis 18: Comparison: Indacaterol Acetate 150 µg vs Placebo; 12 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1619, 95% CI 2-sided [0.0870 to 0.2369]
Statistical Analysis 19: Comparison: Indacaterol Acetate 150 µg vs Placebo; 23 hour 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1249, 95% CI 2-sided [0.0480 to 0.2018]
Statistical Analysis 20: Comparison: Indacaterol Acetate 150 µg vs Placebo; 23 hour 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1546, 95% CI 2-sided [0.0777 to 0.2315]

11. Secondary Outcome: Bronchodilator Effect of Indacaterol Salts Compared to Placebo Measured by FVC (% Predicted)
Description: as for outcome 10
Time Frame: Day 14 of each of the three treatment periods at 5, 15, 30m, 1 2, 3, 4, 8, 12, 23hour.15min and 23hour.45min
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of predicted FVC
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 51 | 52 | 53
Percentage of predicted FVC
  5 min: number analyzed (Participants) | 51 | 52 | 50
  5 min | 90.4 [86.1 to 94.6] | 91.2 [86.9 to 95.4] | 85.3 [81.1 to 89.6]
  15 min: number analyzed (Participants) | 51 | 49 | 51
  15 min | 90.8 [86.6 to 95.1] | 90.7 [86.5 to 95.0] | 84.9 [80.6 to 89.1]
  30 min: number analyzed (Participants) | 51 | 51 | 51
  30 min | 91.6 [87.4 to 95.9] | 91.4 [87.2 to 95.7] | 85.1 [80.8 to 89.3]
  1 hour: number analyzed (Participants) | 51 | 52 | 51
  1 hour | 91.1 [86.8 to 95.3] | 91.1 [86.9 to 95.3] | 85.6 [81.4 to 89.8]
  2 hours: number analyzed (Participants) | 51 | 51 | 51
  2 hours | 90.7 [86.4 to 94.9] | 91.4 [87.1 to 95.6] | 85.9 [81.7 to 90.2]
  4 hours: number analyzed (Participants) | 51 | 51 | 50
  4 hours | 90.5 [86.3 to 94.8] | 91.3 [87.0 to 95.5] | 86.2 [82.0 to 90.5]
  8 hours: number analyzed (Participants) | 49 | 51 | 49
  8 hours | 90.4 [86.1 to 94.6] | 90.3 [86.1 to 94.6] | 85.4 [81.1 to 89.6]
  12 hours: number analyzed (Participants) | 49 | 51 | 48
  12 hours | 88.5 [84.3 to 92.8] | 88.2 [84.0 to 92.5] | 84 [79.8 to 88.3]
  23 hours 15 min: number analyzed (Participants) | 47 | 50 | 41
  23 hours 15 min | 91.5 [87.2 to 95.7] | 89.9 [85.6 to 94.1] | 86.9 [82.6 to 91.2]
  23 hours 45 min: number analyzed (Participants) | 47 | 50 | 41
  23 hours 45 min | 90.6 [86.4 to 94.9] | 90.6 [86.4 to 94.9] | 86.5 [82.3 to 90.8]
Statistical Analysis 1: Comparison: Indacaterol Maleate 150 µg vs Placebo; 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5, 95% CI 2-sided [3.1 to 7.0]
Statistical Analysis 2: Comparison: Indacaterol Maleate 150 µg vs Placebo; 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 6, 95% CI 2-sided [4 to 7.9]
Statistical Analysis 3: Comparison: Indacaterol Maleate 150 µg vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 6.6, 95% CI 2-sided [4.6 to 8.5]
Statistical Analysis 4: Comparison: Indacaterol Maleate 150 µg vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [3.5 to 7.4]
Statistical Analysis 5: Comparison: Indacaterol Maleate 150 µg vs Placebo; 2 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.7, 95% CI 2-sided [2.8 to 6.7]
Statistical Analysis 6: Comparison: Indacaterol Maleate 150 µg vs Placebo; 4 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.3, 95% CI 2-sided [2.3 to 6.3]
Statistical Analysis 7: Comparison: Indacaterol Maleate 150 µg vs Placebo; 8 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5, 95% CI 2-sided [3 to 7]
Statistical Analysis 8: Comparison: Indacaterol Maleate 150 µg vs Placebo; 12 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.5, 95% CI 2-sided [2.5 to 6.5]
Statistical Analysis 9: Comparison: Indacaterol Maleate 150 µg; 23 hour 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [2.6 to 6.7]
Statistical Analysis 10: Comparison: Indacaterol Maleate 150 µg vs Placebo; 23 hour 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [2.0 to 6.2]
Statistical Analysis 11: Comparison: Indacaterol Acetate 150 µg vs Placebo; 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [3.9 to 7.8]
Statistical Analysis 12: Comparison: Indacaterol Acetate 150 µg vs Placebo; 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [3.9 to 7.8]
Statistical Analysis 13: Comparison: Indacaterol Acetate 150 µg vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [4.4 to 8.3]
Statistical Analysis 14: Comparison: Indacaterol Acetate 150 µg vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [3.5 to 7.5]
Statistical Analysis 15: Comparison: Indacaterol Acetate 150 µg vs Placebo; 2 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.5, 95% CI 2-sided [3.5 to 7.4]
Statistical Analysis 16: Comparison: Indacaterol Acetate 150 µg vs Placebo; 4 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [3.1 to 7.0]
Statistical Analysis 17: Comparison: Indacaterol Acetate 150 µg vs Placebo; 8 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [3.0 to 7.0]
Statistical Analysis 18: Comparison: Indacaterol Acetate 150 µg vs Placebo; 12 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [2.2 to 6.2]
Statistical Analysis 19: Comparison: Indacaterol Acetate 150 µg vs Placebo; 23 hour 15 min; Test type: Other; p = 0.004, ANOVA; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [1.0 to 5.0]
Statistical Analysis 20: Comparison: Indacaterol Acetate 150 µg vs Placebo; 23 hour 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 4.1, 95% CI 2-sided [2.1 to 6.1]

12. Secondary Outcome: Bronchodilator Effect of Indacaterol Salts Compared to Placebo Measured by FEV1/FVC
Description: Bronchodilator effect of indacaterol salts compared to placebo in terms of FEV1/FVC at each post dose time point after 14 days. FEV1/FVC ratio is the percentage of the total FVC that is expelled from the lungs during the first second of forced exhalation.
Time Frame: Day 14 of each of the three treatment periods at 5, 15, 30m, 1 2, 3, 4, 8, 12, 23hour.15min and 23hour.45min
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Indacaterol Maleate | Indacaterol Acetate | Placebo
Number analyzed (Participants) | 51 | 52 | 53
Ratio
  5 min: number analyzed (Participants) | 51 | 52 | 50
  5 min | 0.6979 [0.6728 to 0.7230] | 0.6952 [0.6701 to 0.7202] | 0.6729 [0.6478 to 0.6981]
  15 min: number analyzed (Participants) | 51 | 49 | 51
  15 min | 0.7002 [0.6751 to 0.7253] | 0.7017 [0.6766 to 0.7268] | 0.6672 [0.6421 to 0.6923]
  30 min: number analyzed (Participants) | 51 | 51 | 51
  30 min | 0.7012 [0.6761 to 0.7263] | 0.6996 [0.6745 to 0.7246] | 0.6706 [0.6455 to 0.6957]
  1 hour: number analyzed (Participants) | 51 | 52 | 51
  1 hour | 0.7053 [0.6802 to 0.7304] | 0.7007 [0.6757 to 0.7258] | 0.6729 [0.6478 to 0.6980]
  2 hour: number analyzed (Participants) | 51 | 51 | 51
  2 hour | 0.7085 [0.6834 to 0.7336] | 0.7085 [0.6834 to 0.7335] | 0.6747 [0.6496 to 0.6998]
  4 hour: number analyzed (Participants) | 51 | 51 | 50
  4 hour | 0.7057 [0.6806 to 0.7308] | 0.7010 [0.6759 to 0.7261] | 0.6732 [0.6481 to 0.6984]
  8 hour: number analyzed (Participants) | 49 | 51 | 49
  8 hour | 0.6962 [0.6710 to 0.7213] | 0.6967 [0.6716 to 0.7218] | 0.6651 [0.6399 to 0.6902]
  12 hour: number analyzed (Participants) | 49 | 51 | 48
  12 hour | 0.6958 [0.6707 to 0.7210] | 0.6885 [0.6634 to 0.7135] | 0.6599 [0.6348 to 0.6851]
  23 hour 15 min: number analyzed (Participants) | 47 | 50 | 41
  23 hour 15 min | 0.6898 [0.6647 to 0.7150] | 0.6853 [0.6602 to 0.7104] | 0.6572 [0.6320 to 0.6825]
  23 hour 45 min: number analyzed (Participants) | 47 | 50 | 41
  23 hour 45 min | 0.6934 [0.6683 to 0.7186] | 0.6899 [0.6648 to 0.7150] | 0.6633 [0.6381 to 0.6886]
Statistical Analysis 1: Comparison: Indacaterol Maleate vs Placebo; 5 min; Test type: Other; p < .001, ANOVA; Mean Difference (Final Values) = 0.0249, 95% CI 2-sided [0.0139 to 0.0359]
Statistical Analysis 2: Comparison: Indacaterol Maleate vs Placebo; 15 min; Test type: Other; p < .001, ANOVA; Mean Difference (Final Values) = 0.0330, 95% CI 2-sided [0.0220 to 0.0440]
Statistical Analysis 3: Comparison: Indacaterol Maleate vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0306, 95% CI 2-sided [0.0197 to 0.0416]
Statistical Analysis 4: Comparison: Indacaterol Maleate vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0324, 95% CI 2-sided [0.0214 to 0.0434]
Statistical Analysis 5: Comparison: Indacaterol Maleate vs Placebo; 2 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0338, 95% CI 2-sided [0.0228 to 0.0447]
Statistical Analysis 6: Comparison: Indacaterol Maleate vs Placebo; 4 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0325, 95% CI 2-sided [0.0215 to 0.0435]
Statistical Analysis 7: Comparison: Indacaterol Maleate vs Placebo; 8 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0311, 95% CI 2-sided [0.0200 to 0.0422]
Statistical Analysis 8: Comparison: Indacaterol Maleate vs Placebo; 12 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0359, 95% CI 2-sided [0.0248 to 0.0470]
Statistical Analysis 9: Comparison: Indacaterol Maleate vs Placebo; 23 hour 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0326, 95% CI 2-sided [0.0211 to 0.0440]
Statistical Analysis 10: Comparison: Indacaterol Maleate vs Placebo; 23 hour 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0301, 95% CI 2-sided [0.0187 to 0.0415]
Statistical Analysis 11: Comparison: Indacaterol Acetate vs Placebo; 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0222, 95% CI 2-sided [0.0113 to 0.0332]
Statistical Analysis 12: Comparison: Indacaterol Acetate vs Placebo; 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0344, 95% CI 2-sided [0.0234 to 0.0454]
Statistical Analysis 13: Comparison: Indacaterol Acetate vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0290, 95% CI 2-sided [0.0180 to 0.0399]
Statistical Analysis 14: Comparison: Indacaterol Acetate vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0278, 95% CI 2-sided [0.0169 to 0.0387]
Statistical Analysis 15: Comparison: Indacaterol Acetate vs Placebo; 2 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0338, 95% CI 2-sided [0.0228 to 0.0447]
Statistical Analysis 16: Comparison: Indacaterol Acetate vs Placebo; 4 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0278, 95% CI 2-sided [0.0168 to 0.0387]
Statistical Analysis 17: Comparison: Indacaterol Acetate vs Placebo; 8 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0316, 95% CI 2-sided [0.0206 to 0.0426]
Statistical Analysis 18: Comparison: Indacaterol Acetate vs Placebo; 12 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0285, 95% CI 2-sided [0.0175 to 0.0396]
Statistical Analysis 19: Comparison: Indacaterol Acetate vs Placebo; 23 hour 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0281, 95% CI 2-sided [0.0167 to 0.0394]
Statistical Analysis 20: Comparison: Indacaterol Acetate vs Placebo; 23 hour 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.0266, 95% CI 2-sided [0.0152 to 0.0379]

13. Secondary Outcome: Bronchodilator Effect of Indacaterol Salts Compared to Placebo Measured by FEF25-75%
Description: The Forced Expiratory Flow (FEF) 25%-75% measurement describes the amount of air expelled from the lungs during the middle half (25% - 75%) of the forced vital capacity test and is measured using spirometry at each post dose time point after 14 days
Time Frame: Day 14 of each of the three treatment periods at 5, 15, 30m, 1 2, 3, 4, 8, 12, 23hour.15min and 23hour.45min
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters/second
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 51 | 52 | 53
Liters/second
  5 min: number analyzed (Participants) | 51 | 52 | 50
  5 min | 1.6968 [1.4675 to 1.9261] | 1.6918 [1.4628 to 1.9208] | 1.4962 [1.2668 to 1.7256]
  15 min: number analyzed (Participants) | 51 | 49 | 51
  15 min | 1.7454 [1.5160 to 1.9747] | 1.7458 [1.5165 to 1.9751] | 1.4531 [1.2238 to 1.6824]
  30 min: number analyzed (Participants) | 51 | 51 | 51
  30 min | 1.7347 [1.5053 to 1.9640] | 1.7413 [1.5122 to 1.9704] | 1.4690 [1.2397 to 1.6983]
  1 hour: number analyzed (Participants) | 51 | 52 | 51
  1 hour | 1.7715 [1.5422 to 2.0008] | 1.7349 [1.5059 to 1.9640] | 1.4963 [1.2670 to 1.7256]
  2 hour: number analyzed (Participants) | 51 | 51 | 51
  2 hour | 1.7907 [1.5613 to 2.0200] | 1.8074 [1.5782 to 2.0365] | 1.5088 [1.2795 to 1.7381]
  4 hour: number analyzed (Participants) | 51 | 51 | 50
  4 hour | 1.7663 [1.5370 to 1.9956] | 1.7503 [1.5212 to 1.9795] | 1.4843 [1.2549 to 1.7137]
  8 hour: number analyzed (Participants) | 49 | 51 | 49
  8 hour | 1.6755 [1.4460 to 1.9050] | 1.6774 [1.4483 to 1.9066] | 1.4217 [1.1922 to 1.6512]
  12 hour: number analyzed (Participants) | 49 | 51 | 48
  12 hour | 1.6549 [1.4254 to 1.8844] | 1.5849 [1.3557 to 1.8140] | 1.3862 [1.1566 to 1.6158]
  23 hour 15 min: number analyzed (Participants) | 47 | 50 | 41
  23 hour 15 min | 1.6667 [1.4370 to 1.8964] | 1.6257 [1.3965 to 1.8550] | 1.4214 [1.1910 to 1.6518]
  23 hour 45 min: number analyzed (Participants) | 47 | 50 | 41
  23 hour 45 min | 1.6446 [1.4149 to 1.8743] | 1.6580 [1.4288 to 1.8873] | 1.4584 [1.2280 to 1.6866]
Statistical Analysis 1: Comparison: Indacaterol Maleate 150 µg vs Placebo; 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2025, 95% CI 2-sided [0.1059 to 0.2952]
Statistical Analysis 2: Comparison: Indacaterol Maleate 150 µg vs Placebo; 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2923, 95% CI 2-sided [0.1979 to 0.3867]
Statistical Analysis 3: Comparison: Indacaterol Maleate 150 µg vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2657, 95% CI 2-sided [0.1713 to 0.3601]
Statistical Analysis 4: Comparison: Indacaterol Maleate 150 µg vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2752, 95% CI 2-sided [0.1808 to 0.3696]
Statistical Analysis 5: Comparison: Indacaterol Maleate 150 µg vs Placebo; 2 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2819, 95% CI 2-sided [0.1875 to 0.3763]
Statistical Analysis 6: Comparison: Indacaterol Maleate 150 µg vs Placebo; 4 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2820, 95% CI 2-sided [0.1874 to 0.3766]
Statistical Analysis 7: Comparison: Indacaterol Maleate 150 µg vs Placebo; 8 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2538, 95% CI 2-sided [0.1585 to 0.3492]
Statistical Analysis 8: Comparison: Indacaterol Maleate 150 µg vs Placebo; 12 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2687, 95% CI 2-sided [0.1732 to 0.3643]
Statistical Analysis 9: Comparison: Indacaterol Maleate 150 µg vs Placebo; 23 hours 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2453, 95% CI 2-sided [0.1473 to 0.3434]
Statistical Analysis 10: Comparison: Indacaterol Maleate 150 µg vs Placebo; 23 hours 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1862, 95% CI 2-sided [0.0882 to 0.2842]
Statistical Analysis 11: Comparison: Indacaterol Acetate 150 µg vs Placebo; 5 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1956, 95% CI 2-sided [0.1012 to 0.2899]
Statistical Analysis 12: Comparison: Indacaterol Acetate 150 µg vs Placebo; 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2927, 95% CI 2-sided [0.1979 to 0.3875]
Statistical Analysis 13: Comparison: Indacaterol Acetate 150 µg vs Placebo; 30 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2723, 95% CI 2-sided [0.1780 to 0.3667]
Statistical Analysis 14: Comparison: Indacaterol Acetate 150 µg vs Placebo; 1 hour; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2386, 95% CI 2-sided [0.1445 to 0.3328]
Statistical Analysis 15: Comparison: Indacaterol Acetate 150 µg vs Placebo; 2 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2986, 95% CI 2-sided [0.2042 to 0.3930]
Statistical Analysis 16: Comparison: Indacaterol Acetate 150 µg vs Placebo; 4 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2661, 95% CI 2-sided [0.1715 to 0.3607]
Statistical Analysis 17: Comparison: Indacaterol Acetate 150 µg vs Placebo; 8 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2558, 95% CI 2-sided [0.1609 to 0.3506]
Statistical Analysis 18: Comparison: Indacaterol Acetate 150 µg vs Placebo; 12 hours; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1987, 95% CI 2-sided [0.1036 to 0.2938]
Statistical Analysis 19: Comparison: Indacaterol Acetate 150 µg vs Placebo; 23 hours 15 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.2044, 95% CI 2-sided [0.1071 to 0.3017]
Statistical Analysis 20: Comparison: Indacaterol Acetate 150 µg vs Placebo; 23 hours 45 min; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 0.1997, 95% CI 2-sided [0.1023 to 0.2970]

14. Secondary Outcome: Bronchodilator Effect of Indacaterol Salts Compared to Placebo in Standardized FEV1 AUC.
Description: Standardized FEV1 AUC from pre-dose to 4 h post-dose. Evaluated the differences in standardized FEV1 AUC0-4h (L) after 14 days of treatment between indacaterol maleate 150 μg and placebo, and between indacaterol acetate 150 μg and placebo. FEV1 was measured with spirometry conducted according to internationally accepted standards. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time over an entire day (AUC 0-4h)
Time Frame: Pre-dose to 4 hours post-dose on Day 14 of each of the three treatment periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 51 | 52 | 51
Liters | 2.5179 (0.11213) | 2.5151 (0.11205) | 2.2703 (0.11213)
Statistical Analysis 1: Comparison: Indacaterol Maleate 150 µg vs Placebo; Test type: Other; p < .001, ANOVA; Mean Difference (Final Values) = 0.2476, 95% CI 2-sided [0.1857 to 0.3095]
Statistical Analysis 2: Comparison: Indacaterol Acetate 150 µg vs Placebo; Test type: Other; p < .001, ANOVA; Mean Difference (Final Values) = 0.2448, 95% CI 2-sided [0.1830 to 0.3066]
Statistical Analysis 3: Comparison: Indacaterol Maleate 150 µg vs Indacaterol Acetate 150 µg; Test type: Other; ANOVA; Mean Difference (Net) = -0.0028, 95% CI 2-sided [-0.0647 to 0.0590]

15. Secondary Outcome: Rescue Medication Usage
Description: The mean daily number of puffs of rescue medication usage as reported by subjects via diary.
Time Frame: 14 days of treatment for each of the three treatment periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 51 | 52 | 51
Puffs | 1.01 (0.228) | 1.01 (0.227) | 1.43 (0.228)
Statistical Analysis 1: Comparison: Indacaterol Maleate 150 µg vs Placebo; Test type: Other; p = 0.009, ANOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.73 to 0.11]
Statistical Analysis 2: Comparison: Indacaterol Acetate 150 µg vs Placebo; Test type: Other; p = 0.008, ANOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.73 to 0.11]

16. Secondary Outcome: Mean Overall Peak Expiratory Flow (PEF)
Description: A Peak Expiratory Flow (PEF) meter was distributed to patients at Visit 1, to be used to measure PEF twice-daily as directed. During the Screening and Treatment Periods, PEF was measured in the morning and evening every day. the morning PEF was performed within 15 minutes after waking, and the evening PEF approximately 12 hours later. The highest of 3 values was recorded as the daily personal best. The personal best was used to calculate the mean morning PEF and mean evening PEF value collected between assessment Visits LS Mean of change from baseline in mean morning PEF is calculated with the ANOVA model using treatment, stratification group, dosing schedule, gender, center grouping, smoking status, and baseline mean morning PEF as covariates
Time Frame: Days 8 through Day 14 of each of the three treatment periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters/min
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg | Placebo
Number analyzed (Participants) | 51 | 52 | 51
Liters/min | 409.7 (15.06) | 407.6 (15.05) | 376.8 (15.06)
Statistical Analysis 1: Comparison: Indacaterol Maleate 150 µg vs Placebo; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 33.0, 95% CI 2-sided [25.6 to 40.3]
Statistical Analysis 2: Comparison: Indacaterol Acetate 150 µg vs Placebo; Test type: Other; p < 0.001, ANOVA; Mean Difference (Final Values) = 30.8, 95% CI 2-sided [23.5 to 38.2]

ADVERSE EVENTS:
Time Frame: until 30 days after the last Investigational Product (IP) administration
Arm/Group | Indacaterol Maleate 150 µg | Indacaterol Acetate 150 µg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/52 | 0/53
Other Adverse Events (participants affected / at risk) | 14/51 | 7/52 | 9/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol Maleate 150 µg (N=51) | Indacaterol Acetate 150 µg (N=52) | Placebo (N=53)
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol Maleate 150 µg (N=51) | Indacaterol Acetate 150 µg (N=52) | Placebo (N=53)
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT03257995/SAP_000.pdf
  • Study Protocol (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT03257995/Prot_001.pdf